CLINICAL TRIAL: NCT03565419
Title: Application of Smart Glasses During Ultrasound Guided Peripheral Venous Access: a Randomized Controlled Crossover Pilot Study
Brief Title: Use of Smart Glasses for Ultrasound Guided Peripheral Venous Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Joon Min Park, Associate professor, Department of Emergency Medicine, Inje University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2018-04-013
Record Dates: First submitted 2018-05-04; First posted 2018-06-21 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Ultrasonography; Catheterization
MeSH Terms: interventions — Smart Glasses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants conduct the ultrasound-guided peripheral cannulation while they confirm real-time images displayed on the viewer next to the phantom.
- Intervention (Experimental): Participants conduct the ultrasound-guided peripheral cannulation wearing smart glasses. They confirm real-time images displayed on the viewer of smart glasses.
  Interventions: Device: Smart glasses

INTERVENTIONS:
Device: Smart glasses — Participants confirm the real-time ultrasound image displayed on the viewer of smart glasses.
  Arms: Intervention

SUMMARY:
Investigators aimed to explore the feasibility of smart glasses connected to a wireless ultrasound transducer for the peripheral venous access. Residents who have basic skills of ultrasound guided procedure participate in the simulation. Each participant plays the following two roles for ultrasound guided peripheral venous access; ultrasound guided peripheral venous access with and without wearing smart glasses. The order of performing two roles is determined by a randomized process and the gap between two roles are five days. The primary outcome is the time of successful blood aspiration, and secondary outcomes are first time success rate, the number of skin puncture, the number of needle redirection, the number of head movement, and subjective difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Doctors who have basic skill for the ultrasound guided procedures and agree to participate the simulation

Exclusion Criteria:

* Doctors who do not agree to participate the simulation
* Doctors who do not have basic skill for the ultrasound guided procedures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
time for successful blood aspiration | up to 1 month
  duration from application of probe to successful aspiration

SECONDARY OUTCOMES:
first time success rate | up to 1 month
  chance for successful aspiration within 90 seconds
number of skin puncture | up to 1 month
  number of skin puncture during ultrasound guided venous access
number of needle redirection | up to 1 month
  number of needle redirection during ultrasound guided venous access
number of head movement | up to 1 month
  number of participant's head movement during ultrasound guided venous access
subjective difficulty of procedure | up to 1 month
  measuring subjective difficulty with the 100mm VAS (0: easy, 100: difficult)

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Ilsan Paik Hospital, Goyang-si, South Korea

IPD SHARING:
Plan to Share IPD: No